CLINICAL TRIAL: NCT00540358
Title: A Phase 2, Multi-center, Open-Label, Randomized Trial of Gemcitabine/ Carboplatin, With or Without BSI-201, in Patients With ER, PR and HER2-negative Metastatic Breast Cancer
Brief Title: A Phase 2 Trial of Standard Chemotherapy, With or Without BSI-201, in Patients With Triple Negative Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: BiPar Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCD11485; 20070102 (Other: BiPar)
Expanded Access: NCT01130259 (No longer available)
Record Dates: First submitted 2007-10-04; First posted 2007-10-08 (Estimated); Last update posted 2012-12-28 (Estimated); Status verified 2012-12

CONDITIONS: Breast Cancer
Keywords: Triple negative breast cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Gemcitabine; Carboplatin; iniparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm G/C (Active Comparator): Standard chemotherapy with gemcitabine/carboplatin on Days 1 and 8 of 21-day cycle(s)
  Interventions: Drug: gemcitabine/carboplatin
- Arm G/C/I (Experimental): Standard chemotherapy with gemcitabine/carboplatin on Days 1 and 8, plus iniparib on Days 1, 4, 8, and 11 of 21-day cycle(s)
  Interventions: Drug: gemcitabine/carboplatin; Drug: iniparib

INTERVENTIONS:
Drug: gemcitabine/carboplatin — Gemcitabine and carboplatin administered according to instructions in the package inserts.
Drug: iniparib — Body weight adjusted dose
  1 hour intravenous infusion
  Other Names: BSI-201; SAR240550
  Arms: Arm G/C/I

SUMMARY:
The purpose of this clinical trial was to determine whether combining iniparib (BSI-201) with standard chemotherapy in estrogen receptor (ER)-negative, progesterone receptor (PR)-negative, and human epidermal growth factor receptor 2 (HER2) negative metastatic breast cancer patients improve clinical benefit compared to treatment with standard chemotherapy alone.

Based on data generated by BiPar/Sanofi, it was concluded that iniparib does not possess characteristics typical of the poly (ADP-ribose) polymerase (PARP) inhibitor class. The exact mechanism has not yet been fully elucidated, however based on experiments on tumor cells performed in the laboratory, iniparib is a novel investigational anti-cancer agent that induces gamma-H2AX (a marker of DNA damage) in tumor cell lines, induces cell cycle arrest in the G2/M phase in tumor cell lines, and potentiates the cell cycle effects of DNA damaging modalities in tumor cell lines. Investigations into potential targets of iniparib and its metabolites are ongoing.

DETAILED DESCRIPTION:
Patients were treated until disease progression, unacceptable toxicity, Investigator's decision to discontinue, or withdrawal of consent. After treatment discontinuation, all patients were evaluated every 90 days after last dose of gemcitabine/carboplatin with or without iniparib, for up to 3 years or death or end of study, which ever occurred first.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age;
* Metastatic breast cancer (Stage IV) with measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) criteria;
* 0-2 prior chemotherapy regimens in the metastatic setting;
* Histologically documented (either primary or metastatic site) breast cancer that was ER-negative, PR-negative, and HER-2 nonoverexpressing by immunohistochemistry (0,1) or non-gene amplification by fluorescence in situ hybridization (FISH);
* Completion of prior chemotherapy at least 2 weeks prior to trial entry and recovery from toxicity of prior chemotherapy;
* Radiation therapy must have been completed at least 2 weeks prior to trial entry, and radiated lesions may not have served as measurable disease;
* Patient may have had central nervous system (CNS) metastases if he/she did not require steroids, whole brain radiation therapy (XRT), gamma/cyber knife, and brain metastases were clinically stable without symptomatic progression;
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1;
* Adequate organ function defined as: absolute neutrophil count (ANC)≥1,500/mm3, platelets ≥100,000/mm3, creatinine clearance >50mL/min, ALT and AST <2.5 x upper limit of normal (ULN) (or <5 x ULN in case of liver metastases); total bilirubin <1.5 mg/dL.
* Tissue block (primary or metastatic) available for PARP and PG studies was recommended, although its absence did not exclude subjects from participating;
* Woman of child bearing potential must have had documented negative pregnancy test within two weeks of trial entry and agreed to acceptable birth control during the duration of the trial therapy;
* Signed, IRB approved written informed consent.

Exclusion Criteria:

* Lesions identifiable only by positron emission tomography (PET);
* Prior treatment with gemcitabine, carboplatin, cisplatin or iniparib;
* Major medical conditions that might have affected trial participation (uncontrolled pulmonary, renal, or hepatic dysfunction, uncontrolled infection);
* Significant history of uncontrolled cardiac disease; i.e. uncontrolled hypertension, unstable angina, recent myocardial infarction (within prior 6 months), uncontrolled congestive heart failure, and cardiomyopathy that was either symptomatic or asymptomatic but with decreased ejection fraction <45%;
* Other significant comorbid condition which the investigator felt might compromise effective and safe participation in the trial;
* Patient enrolled in another investigational device or drug trial, or was receiving other investigational agents;
* Concurrent or prior (within 7 days of trial day 1) anticoagulation therapy (low dose for port maintenance allowed);
* Concurrent radiation therapy was not permitted throughout the course of the trial;
* Inability to comply with the requirements of the trial;
* Pregnant or lactating woman;
* Leptomeningeal disease or brain metastases requiring steroids or other therapeutic intervention.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2007-10; Primary Completion 2009-11 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Clinical benefit rate | until cut-off date established so that all patients were evaluable for primary outcome measure
  Clinical benefit rate was defined as the percentage of patients with complete response, partial response or stable disease ≥6 months.

SECONDARY OUTCOMES:
Objective response rate | until cut-off date established so that all patients were evaluable for primary outcome measure
  Objective response rate was defined as the percentage of patients with confirmed partial response or complete response
Progression-free survival | until cut-off date established so that all patients were evaluable for primary outcome measure
  Progression-free survival was defined as the time interval from the date of randomization to the date of disease progression or the date of death due to any cause, whichever came first.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (18):
- United States (18):
  - Research Site, Birmingham, Alabama
  - Research Site, Denver, Colorado
  - Research Site, Torrington, Connecticut
  - Research Site, Ocoee, Florida
  - Research Site, Indianapolis, Indiana
  - Research Site, Overland Park, Kansas
  - Research Site, Henderson, Nevada
  - Research Site, Hooksett, New Hampshire
  - Research Site, Raleigh, North Carolina
  - Research Site, Bedford, Texas
  - Research Site, Dallas, Texas
  - Research Site, El Paso, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, Tyler, Texas
  - Research Site, Fairfax, Virginia
  - Research Site, Vancouver, Washington
  - Research Site, Yakima, Washington

REFERENCES:
- [Result] O'Shaughnessy J, Osborne C, Pippen JE, Yoffe M, Patt D, Rocha C, Koo IC, Sherman BM, Bradley C. Iniparib plus chemotherapy in metastatic triple-negative breast cancer. N Engl J Med. 2011 Jan 20;364(3):205-14. doi: 10.1056/NEJMoa1011418. Epub 2011 Jan 5. PMID 21208101